CLINICAL TRIAL: NCT03418142
Title: Research Evaluating the EffectiVeness of Adding an Internet-Based Self-Management Intervention to Usual Care in the Treatment of Borderline Personality Disorder - REVISIT BPD
Brief Title: Evaluating an Internet-Based Self-Management Intervention for Borderline
Acronym: REVISIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gaia AG (Industry)
Collaborators: University of Luebeck (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REVISIT-BPD Trial
Record Dates: First submitted 2018-01-23; First posted 2018-02-01 (Actual); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: Borderline Personality Disorder
MeSH Terms: conditions — Borderline Personality Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Priovi (Experimental): Priovi is an Internet-administered intervention for people with BPD.
  Interventions: Behavioral: Priovi; Other: CAU
- Care-as-Usual (CAU) / wait list (Active Comparator): Additionaly, they will be informed about helpful and free available online self-help-proposals for BPD patients immediately after randomization.
  Interventions: Other: CAU

INTERVENTIONS:
Behavioral: Priovi — Priovi is an Internet intervention for people with BPD. Content is continuously adapted to patients' concerns and needs. Priovi is a comprehensive program, which is conceptually and substantially based on the schema therapeutic approach used in BPD patients. It contains interactive dialogues that can be accessed via computer or smartphone, illustrations, audios and motivating text messages. Techniques to cope with borderline symptoms (e.g., psychoeducation about modes, schemas and basic emotional needs in addition to relevant strategies to weaken, reduce and/or heal maladaptive schemas and modes) are conveyed in interactive sequences that are accompanied by audio recordings, illustrations, and worksheets. Patients are also prompted to regularly complete brief symptom severity self-monitoring questionnaires. Optional daily text messages with motivational content accompany the program. The program can be accessed for 365 days after registration.
  Arms: Priovi
Other: CAU — Care as Usual: In the CAU/wait list control group, participants are free to continue to engage with any treatment they require (i.e., CAU). However, they will receive access to Priovi after 12 months post-baseline (i.e., wait list with respect to Priovi access).

SUMMARY:
The trial aims to evaluate the effectiveness of a novel internet intervention (Priovi), which was designed to introduce relevant schema therapy techniques to Persons with Borderline Personality Disorder (BPD). Therefore, 200 people with BPD will be recruited and randomized to two groups: (1) a control group, in which they may engage with any BPD treatment (Care-as-Usual, CAU) and receive access to Priovi after a delay of 12 months (i.e., CAU/wait list control group), or (2) to a treatment group that immediately receives 12-month access to Priovi and may also use CAU. The primary outcome measure is the score of the Borderline Personality Disorder Severity Index (BPDSI), collected at three, six and 12 month post-baseline.

DETAILED DESCRIPTION:
In the treatment of psychological disorders, web-based self-help programs can be very helpful, especially when combined with psychotherapy. However, up to this point, there are no respective programs for patients with Borderline Personality Disorder (BPD), although this disorder is associated with severe personal suffering and requires time-consuming therapy, which, in many cases, cannot be provided, due to the lack of therapeutic supply.

In this study, treatment effects of the web-based self-help program Priovi on BPD symptom severity when added to treatment as usual will be investigated. Priovi is a comprehensive program, which is conceptually and substantially based on the schema therapeutic approach used in BPD patients. It contains interactive dialogues that can be accessed via computer or smartphone, illustrations, audios and motivating text messages.

After a phone pre-screen and a diagnostic evaluation conducted by a psychiatrist, 200 patients suffering from BPD will be randomized into either the intervention group or into the waitlist control group. Priovi's duration of use is one year, measuring points will be determined before beginning of treatment (T0) as well as after 3 (T1), 6 (T2), 9 (T3) and 12 months (T4). The primary outcome variable will be the score of the Borderline Personality Disorder Severity Index (BPDSI), a highly reliable external assessment tool measuring BPD severity. Secondary outcome variables will be BPD symptom severity (as assessed by self-ratings), symptom severity of depression and anxiety as well as quality of life. The study will be collaboratively conducted by the University of Lübeck and the GAIA AG in Hamburg.

In this study, Priovi for BPD patients will be tested in a randomized controlled trial. It will be used as add-on therapy combined with any guideline therapy available to the respective patients. In doing so, the following hypothesis will be investigated: Compared to patients, who exclusively receive treatment as usual, the additional use of the self-help program in question will lead to a stronger decrease in BPD symptom severity.

ELIGIBILITY:
Inclusion Criteria:

* Psychiatric diagnosis of BPD
* BPDSI score of 15 or higher
* Informed consent
* German language proficiency
* Willingness to participate in diagnostic and follow-up assessments as well as to see a -
* Psychiatrist for validation of diagnosis
* 18 years or older

Exclusion Criteria:

* Psychotic disorder
* Primary psychiatric diagnosis of an addictive disorder
* Schizotypal personality disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2018-01-29 (Actual); Primary Completion 2020-01-29 (Actual); Study Completion 2020-01-29 (Actual)

PRIMARY OUTCOMES:
Score of the Borderline Personality Disorder Severity Index (BPDSI) - The BPDSI is a semi-structured interview assessing the frequency and severity of manifestations of borderline personality disorder (BPD) during the last three months. | Changes from baseline to 3, 6 and 12 months
  Semi-structured interview assessing BPD symptom frequency and severity

SECONDARY OUTCOMES:
Severity of depressive symptoms, measured by Patient Health Questionnaire - 9 items (PHQ-9) | Changes from baseline to 3, 6, 9 and 12 months.
  Self-report depression symptom severity measure.
  Nine items, each of which is scored 0 to 3, providing a 0 to 27 severity score.
  Depression Severity: 0-4 none, 5-9 mild, 10-14 moderate, 15-19 moderately severe, 20-27 severe.
GAD-7 (Generalized Anxiety Disorder Questionnaire) | Changes from baseline to 3, 6, 9 and 12 months.
  Self-report anxiety symptom severity measure.
  Seven items, each of which is scored 0 to 3, providing a 0 to 21 severity score.
  Anxiety Severity: 0-4 none, 5-9 mild, 10-14 moderate, 15-21 severe.
EQ-5D (standardized instrument developed by the EuroQol Group as a measure of health-related quality of life.) | Changes from baseline to 3, 6, 9 and 12 months.
  Self-report measure of quality of life symptoms.
BPD-Checklist short (Borderline personality Disorder Checklist short) | Changes from baseline to 3, 6, 9 and 12 months.
  Self-report measure of BPD symptoms.
2 Items of CIUS-Long-brief (Compulsive Internet Use Scale) | Assessed at 3, 6, 9 and 12 months.
  Adapted self-report measure assessing potential compulsive internet use.
  two items, each of which is scored 1 to 5, providing a 2 to 10 severity score with higher values representing a worse outcome
NEQ (negative effects questionnaire) | Assessed at baseline, 3, 6, 9 and 12 months.
  Self-report measure of potential negative effects of the treatment.
  qualitative measure.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Philipp Klein, Dr. med., Principal Investigator — University of Lübeck, Zentrum für Integrative Psychiatrie ZiP gGmbH
Locations (1):
- Gaia AG, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual participant data shall be made available upon request for projects such as meta-analyses after completion of the study

REFERENCES:
- [Derived] Klein JP, Hauer-von Mauschwitz A, Berger T, Fassbinder E, Mayer J, Borgwardt S, Wellhofer B, Schweiger U, Jacob G. Effectiveness and safety of the adjunctive use of an internet-based self-management intervention for borderline personality disorder in addition to care as usual: results from a randomised controlled trial. BMJ Open. 2021 Sep 8;11(9):e047771. doi: 10.1136/bmjopen-2020-047771. PMID 34497078
- [Derived] Storebo OJ, Stoffers-Winterling JM, Vollm BA, Kongerslev MT, Mattivi JT, Jorgensen MS, Faltinsen E, Todorovac A, Sales CP, Callesen HE, Lieb K, Simonsen E. Psychological therapies for people with borderline personality disorder. Cochrane Database Syst Rev. 2020 May 4;5(5):CD012955. doi: 10.1002/14651858.CD012955.pub2. PMID 32368793
- [Derived] Klein JP, Hauer A, Berger T, Fassbinder E, Schweiger U, Jacob G. Protocol for the REVISIT-BPD Trial, a Randomized Controlled Trial Testing the Effectiveness of an Internet-Based Self-Management Intervention in the Treatment of Borderline Personality Disorder (BPD). Front Psychiatry. 2018 Sep 21;9:439. doi: 10.3389/fpsyt.2018.00439. eCollection 2018. PMID 30298024